CLINICAL TRIAL: NCT07133646
Title: Effect of Rib Mobilization and Diaphragm Release Techniques in Patients With Non-Specific Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ahmed Abd El hady El Fahl,ph.d, Assisstant professor, MTI University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB # 28/7/2024-2025
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RMT and DRT(Rib Mobilization Technique and Diaphragm Release Technique) (Experimental): Rib Mobilization Technique and Diaphragm Release Technique(In the seated position, the participants remained seated on the stretcher, keeping the feet on the floor, while the therapist stood in front of him or her. The participant's head (frontal region) was positioned over his or her overlapping arms, which were placed on the therapist's trunk )
  Interventions: Other: Rib Mobilization Technique and Diaphragm Release Technique; Other: Diaphragm Release Technique
- DRT(Diaphragm Release Technique) (Experimental): Diaphragm Release Technique:The DRT was performed according to the protocol described by Rocha et al.13 In this protocol, the participant remains in the supine position so that the therapist is able to maintain manual contact with the bottom edge of the rib cage
  Interventions: Other: Diaphragm Release Technique
- control (No Intervention): No intervention

INTERVENTIONS:
Other: Rib Mobilization Technique and Diaphragm Release Technique — The RMT, adapted from Henderson et al10 and Abdelaal et al,15 was carried out in 2 different participant positions: supine and seated. In the supine position, the therapist was placed next to the participant and positioned the last 4 fingertips of both hands at the rib angles. The therapist mobilized the costal angles in the postero anterior direction accompanying the participant's normal inspiration The movement was performed in 2 series of 10 respiratory cycles in each hemi thorax, with a 1-minute interval between sets.
  Arms: RMT and DRT(Rib Mobilization Technique and Diaphragm Release Technique)
Other: Diaphragm Release Technique — The DRT was performed according to the protocol described by Rocha et al.13 In this protocol, the participant remains in the supine position so that the therapist is able to maintain manual contact with the bottom edge of the rib cage. During inspiration, the therapist exerts traction after the natural rib-cage movement, then deepens the manual contact and maintains the resistance exerted in the previous phase throughout exhalation. The technique was applied in 2 series of 10 deep respiratory cycles, with a 1-minute interval between the series, under the therapist's verbal command.
  Arms: DRT(Diaphragm Release Technique); RMT and DRT(Rib Mobilization Technique and Diaphragm Release Technique)

SUMMARY:
Rib mobilization is a therapeutic technique aimed at enhancing the mobility of the ribcage, which can have a significant impact on neck pain, even when the pain is classified as non-specific. The ribcage plays a crucial role in maintaining the alignment and posture of the upper body, including the neck. When the ribs are restricted or misaligned, it can lead to compensatory movements and increased strain on the cervical spine, contributing to neck pain. By mobilizing the ribs, we can restore their natural movement, which in turn can release tension in the surrounding musculature and improve the overall biomechanics of the thoracic and cervical regions. This approach not only addresses the immediate symptoms of neck pain but also targets the underlying structural issues that may perpetuate discomfort.

DETAILED DESCRIPTION:
The diaphragm is a major muscle involved in respiration, but its function extends beyond just breathing. It acts as a core stabilizer and influences the mechanics of the thoracic and cervical areas. Tension or dysfunction in the diaphragm can lead to altered breathing patterns and increased tension in the neck and shoulders, exacerbating non-specific neck pain. Releasing the diaphragm can improve respiratory efficiency and reduce undue stress on the neck. This release helps in re-establishing a more natural breathing pattern, which can alleviate pain and improve overall posture. Additionally, by addressing the diaphragm, we can indirectly affect the autonomic nervous system, promoting relaxation and reducing stress, which are often contributing factors to chronic pain syndromes.

An integrated approach that combines rib mobilization and diaphragm release can be particularly effective for managing non-specific neck pain. This method not only targets the symptoms but also addresses the root causes of neck discomfort. By improving rib and diaphragm function, we enhance the body's ability to maintain proper posture and reduce compensatory strain on the neck. This holistic treatment strategy is essential because it recognizes the interconnectedness of the body's musculoskeletal and respiratory systems. Furthermore, this approach empowers patients by providing them with a deeper understanding of their body mechanics and encouraging active participation in their rehabilitation process. Through this combination of manual therapy techniques, patients are likely to experience improved mobility, reduced pain, and a greater sense of well-being.

ELIGIBILITY:
Inclusion Criteria:

* Neurological tests will be negative
* Both genders having age between 20 to 45 years
* Participants should have primary complaint of neck pain
* Neck Disability Index (NDI) score of 20% or greater (i.e. 10 points or greater on a 0 to 50 scale)
* A pain intensity of ≥4 on the 10-point Numerical Pain Rating Scale (NPRS)

Exclusion Criteria:

* First and second rib fracture and dislocation
* Past surgical history of cervical and thoracic region
* Thoracic Outlet syndrome and cervical radiculopathy
* Congenital anomalies of spine and ribs

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) | at baseline and at 8 weeks
  The Numerical Pain Rating Scale (NPRS) is a subjective measure used to assess the intensity of neck pain in individuals. Patients are asked to rate their pain on a scale from 0 to 10, where 0 represents "no pain" and 10 signifies "the worst possible pain." This simple tool provides a quantitative measure of pain, enabling healthcare providers to evaluate the severity of the patient's condition and monitor changes over time. The NPRS is widely used due to its ease of application and effectiveness in capturing patient-reported pain intensity
Neck range of motion (ROM) | at baseline and at 8 weeks
  A goniometer is an instrument used to measure the range of motion (ROM) of the neck. It is an essential tool for evaluating the flexibility and mobility of the cervical spine. During the assessment, the goniometer is aligned with specific anatomical landmarks to measure the angles of neck flexion, extension, lateral flexion, and rotation. This objective data is crucial for identifying limitations in neck movement, which could contribute to pain and functional impairment. The goniometer is considered reliable and valid for assessing cervical ROM in clinical settings

SECONDARY OUTCOMES:
Neck flexor Muscle Endurance Test | at baseline and at 8 weeks
  The muscle endurance test for the neck involves assessing the endurance of neck muscles by measuring the duration a patient can maintain a certain position against gravity. A common method is the neck flexor endurance test, where the patient lies supine and holds their head off the table. The time held without compensatory movements is recorded using a stopwatch. This test helps in identifying muscle weakness or endurance deficits that may contribute to neck pain. Muscle endurance is a critical component of neck function, and its assessment is important for tailoring rehabilitation programs
Neck Disability Index | at baseline and at 8 weeks
  The Neck Disability Index (NDI) is a self-reported questionnaire designed to measure the impact of neck pain on daily activities and overall quality of life. It consists of 10 items addressing pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreation. Each item is scored from 0 to 5, with higher scores indicating greater disability. The NDI is a validated tool widely used in both clinical and research settings to assess the functional status of individuals with neck pain and to monitor treatment outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy ,Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No